CLINICAL TRIAL: NCT01343186
Title: A Single-centre, Randomised, Positive-controlled, Single-dose, Dose-escalation Study to Assess Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Ypeginterferon Alfa-2a in Healthy Subjects
Brief Title: Safety, Tolerability, Pharmacokinetics and Pharmacodynamics Assessment of Ypeginterferon Alfa-2a in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Xiamen Amoytop Biotech Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple
Other Study IDs: TB1012IFN
Record Dates: First submitted 2011-04-24; First posted 2011-04-27 (Estimated); Last update posted 2012-01-31 (Estimated); Status verified 2010-12

CONDITIONS: Healthy Subjects
Keywords: Peginterferon; Healthy subject; Pharmacokinetics; Pharmacodynamics; Safety
MeSH Terms: interventions — peginterferon alfa-2a

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Arm 1 (Other)
  Interventions: Drug: Peginterferon alfa
- Arm 2 (Other)
  Interventions: Drug: Peginterferon alfa 2a
- Arm 3 (Other)
  Interventions: Drug: Peginterferon alfa-2a
- Arm 4 (Other)
  Interventions: Drug: Peginterferon alfa-2a

INTERVENTIONS:
Drug: Peginterferon alfa — s,c, 45mcg of Ypeginterferon alfa-2a
  Arms: Arm 1
Drug: Peginterferon alfa 2a — s,c, 90mcg of Ypeginterferon alfa-2a or 180mcg of Pegasys.
  Arms: Arm 2
Drug: Peginterferon alfa-2a — s,c, 180mcg of Ypeginterferon alfa-2a or 180mcg of Pegasys.
  Arms: Arm 3
Drug: Peginterferon alfa-2a — s,c, 270mcg of Ypeginterferon alfa-2a or 180mcg of Pegasys.
  Arms: Arm 4

SUMMARY:
This study is aimed to study the pharmacokinetic characteristics(e.g. AUC, Cmax, Tmax) of Ypeginterferon alfa-2a and interferon biomarkers(e.g. 2,5-OAS, neopterin) after single dose at different levels.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects
* Age between 18 and 45, inclusive
* Body mass index(BMI)between 19 and 26, inclusive
* Sign informed consent

Exclusion Criteria:

* Women of pregnant or lactation
* Known hypersensitivity to interferon or any other components of the study drug
* History of mental disease or genetic disease
* History of diabetes mellitus, thyroid disease, cancer, autoimmune disease, organ transplant
* Significant disease in heart, liver, kidney, lung or any other major organs
* Alcoholic, smokers or drug abusers
* Blood donation, or massive blood loss due to injury or surgery within 3 months
* Other conditions which in the opinion of the investigator preclude enrollment into the study

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 39 (Actual)
Dates: Start 2011-01; Primary Completion 2011-05 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Measuring interferon levels in blood samples | from 0 to 408 hours following injection
Different blood interferon biomarkers (such as 2,5-OAS, neopterin) | from 0 to 408 hours following injection

SECONDARY OUTCOMES:
Adverse events | up to 3 weeks following injection
Anti-interferon antibody | baseline and week 2 after injection

CONTACTS AND LOCATIONS:
Overall Officials: Wei Zhenman, Ph.D, Principal Investigator — Beijing 302 Hospital
Locations (1):
- 302 Military Hospital of China, Beijing, China